CLINICAL TRIAL: NCT01253161
Title: Phase II Study of Pasireotide LAR in Patients With Metastatic Neuroendocrine Carcinomas
Brief Title: Study of Pasireotide Long Acting Release (LAR) in Patients With Metastatic Neuroendocrine Tumors (NETs)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis Pharmaceuticals (Industry); RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16438; CSOM230DUS23T (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2010-11-30; First posted 2010-12-03 (Estimated); Results first posted 2022-01-18 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Neuroendocrine Tumors; Carcinoid Tumors
Keywords: advanced; metastatic; unresectable; carcinoma; gastrointestinal tract; lungs; colon; liver; rectum; small intestine; stomach; pancreatic
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor; Neoplasm Metastasis; Carcinoma | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pasireotide LAR Treatment (Experimental): The investigational drug used in this study is pasireotide long acting release (LAR) 60 mg.
  Interventions: Drug: Pasireotide Long Acting Release (LAR)

INTERVENTIONS:
Drug: Pasireotide Long Acting Release (LAR) — Pasireotide will be administered as an intramuscular injection at the beginning of every cycle which is defined as 28 days (+/- 3 days). Study treatment should begin within 14 days following enrollment into the study and continue until disease progression, unacceptable toxicity, or withdrawal of consent.
  Other Names: SOM 230

SUMMARY:
The goal of this clinical research study is to learn if the study drug, Pasireotide LAR can shrink or slow the growth of Metastatic Neuroendocrine Carcinomas. The safety of this drug will also be studied. The patient's physical state, changes in the size of the tumor, and laboratory findings taken while on-study will help us decide if Pasireotide LAR is safe and effective.

DETAILED DESCRIPTION:
This is a multi-institutional, prospective phase II open-label trial.

The investigational drug used in this study is pasireotide LAR 60 mg. Pasireotide will be administered as an intramuscular injection at the beginning of every cycle which is defined as 28 days (+/- 3 days). Study treatment should begin within 14 days following enrollment into the study and continue until disease progression, unacceptable toxicity, or withdrawal of consent. Safety and efficacy will be assessed throughout the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Locally unresectable or metastatic carcinoid or pancreatic neuroendocrine tumors
* Tumors must be considered well or moderately differentiated (or low to intermediate grade). Patients with poorly differentiated neuroendocrine carcinomas or small cell carcinomas are excluded from the study.
* No prior systemic antineoplastic neuroendocrine tumor treatment (including prior somatostatin analogs). However patients who have received a short course of subcutaneous (SQ) octreotide (<10 days) in the past are eligible if > 1 week has elapsed from their last octreotide injection.
* Minimum of four weeks since any major surgery
* Measureable disease by Response Evaluation Criteria in Solid Tumors (RECIST)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Life expectancy 12 weeks or more
* Adequate bone marrow function as shown by: absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L, Platelets ≥ 75 x 10^9/L, hemoglobin (Hgb) > 8 g/dL
* Adequate liver function as shown by: serum bilirubin ≤ 2.0 x upper limit of normal (ULN), and serum transaminases activity ≤ 2 x ULN, with the exception of serum transaminases (< 3 x ULN) if the patient has liver metastases
* Adequate renal function as shown by serum creatinine ≤ 2.0 x ULN
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. Note: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 14 days of the administration of the first study treatment. Women must not be lactating. Both men and WOCBP must be advised of the importance of using effective birth control measures during the course of the study.
* Signed informed consent to participate in the study must be obtained from patients after they have been fully informed of the nature and potential risks by the investigator (or his/her designee) with the aid of written information.

Exclusion Criteria:

* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Patients with prior or concurrent malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, or other adequately treated in situ cancer, or any other cancer from which the patient has been disease free for 5 years
* Patients with uncontrolled diabetes mellitus or a fasting plasma glucose > 1.5 ULN or glycosylated hemoglobin (HbA1c) >8%. Note: At the principle investigator's discretion, non-eligible patients can be re-screened after adequate medical therapy has been instituted.
* Patients with symptomatic cholelithiasis
* Patients who have congestive heart failure: New York Heart Association (NYHA) Class III or IV, unstable angina, or a history of acute myocardial infarction within the 6 months preceding enrollment
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * Severely impaired lung function
  * Any active (acute or chronic) or uncontrolled infection/ disorders
  * Nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy
* Known hypersensitivity to somatostatin analogues or any component of the pasireotide LAR formulation
* Corrected QT interval (QTcF) of >470 msec on screening Electrocardiogram (ECG)
* Risk factors for Torsades de Pointes such as cardiac failure, clinically significant/symptomatic bradycardia
* Clinically significant hypokalemia or hypomagnesemia that are not correctable
* History of sustained ventricular tachycardia, ventricular fibrillation, advanced heart block, or idiopathic syncope thought to be related to ventricular arrhythmia
* Concomitant medication(s) known to increase the QT interval
* History of noncompliance to medical regimens or unwillingness to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-02-01 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2023-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Strosberg, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - Stanford Cancer Institute, Stanford, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida

REFERENCES:
- [Derived] Cives M, Kunz PL, Morse B, Coppola D, Schell MJ, Campos T, Nguyen PT, Nandoskar P, Khandelwal V, Strosberg JR. Phase II clinical trial of pasireotide long-acting repeatable in patients with metastatic neuroendocrine tumors. Endocr Relat Cancer. 2015 Feb;22(1):1-9. doi: 10.1530/ERC-14-0360. Epub 2014 Nov 6. PMID 25376618

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pasireotide LAR Treatment
Started | 29
Completed | 28
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pasireotide LAR Treatment
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 23
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) at One Year
Description: PFS: Defined as the time from the date of first study treatment to the date of the first documented disease progression, by Response Evaluation Criteria in Solid Tumors (RECIST 1.0) guidelines, or death due to any cause. Progressive Disease (PD): at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 12 months
Population: Evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pasireotide LAR Treatment
Number analyzed (Participants) | 28
months | 11 [7.6 to 16]

2. Secondary Outcome: Overall Radiographic Response Rate (ORR)
Description: Complete response (CR): complete disappearance of all target lesions, confirmed by repeat assessments at no less than 4 weeks after the criteria for response are first met. Partial response (PR): at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. This must be confirmed by repeat assessment at no less than 4 weeks after the criteria for response are first met. Stable Disease (SD): neither sufficient decrease to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter since the treatment started.
Time Frame: Up to 48 months
Population: evaluable participants
Measure: Number; unit: percentage of participants
Arm/Group | Pasireotide LAR Treatment
Number analyzed (Participants) | 28
percentage of participants
  Partial Response | 4
  Stable Disease | 60
  Progressive Disease | 36

3. Secondary Outcome: Adverse Events Possibly Related to Study Treatment
Description: Adverse Events (AEs) and Serious Adverse Events (SAEs) will be evaluated continuously throughout the study. Safety and tolerability will be assessed according to the NIH/NCI Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0).
Time Frame: Up to 48 months
Population: All participants who received at least one dose of study drug
Measure: Number; unit: events
Arm/Group | Pasireotide LAR Treatment
Number analyzed (Participants) | 29
events | 42

ADVERSE EVENTS:
Time Frame: Adverse events collected for 28 days after last dose of study drug, up to 60 months.
Arm/Group | Pasireotide LAR Treatment
All-Cause Mortality (participants affected / at risk) | 6/29
Serious Adverse Events (participants affected / at risk) | 12/29
Other Adverse Events (participants affected / at risk) | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pasireotide LAR Treatment (N=29)
Platelet count decreased (Investigations) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Cardiac Disorders - Other (Cardiac disorders) | 1 (1)
Dueodenal obstruction (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — Perirectal abcess
Nausea (Gastrointestinal disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1) — Urinary tract infection
Creatinine increased (Investigations) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Ileal obstruction (Gastrointestinal disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pasireotide LAR Treatment (N=29)
Hyperglycemia (Metabolism and nutrition disorders) | 24 (147)
Anorexia (Metabolism and nutrition disorders) | 4 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (14)
Hyponatremia (Metabolism and nutrition disorders) | 2 (12)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (5)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 11 (13)
Abdominal pain (Gastrointestinal disorders) | 9 (17)
Constipation (Gastrointestinal disorders) | 6 (7)
Nausea (Gastrointestinal disorders) | 5 (6)
Vomiting (Gastrointestinal disorders) | 5 (6)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 4 (4)
Bloating (Gastrointestinal disorders) | 2 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 12 (19)
Edema limbs (General disorders) | 4 (4)
Pain (General disorders) | 3 (3)
Chills (General disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (General disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 3 (4)
Alanine aminotransferase increased (Investigations) | 2 (8)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 2 (5)
Weight loss (Investigations) | 2 (3)
Blood bilirubin increased (Investigations) | 1 (1)
Investigations - Other (Investigations) | 1 (1)
Pancreatic enzymes decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (3)
Weight gain (Investigations) | 1 (2)
Hypertension (Vascular disorders) | 8 (30)
Flushing (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (7)
Dizziness (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Blurred vision (Eye disorders) | 2 (2)
Eye disorders - Other (Eye disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (6)
Cardiac disorders - Other (Cardiac disorders) | 2 (3)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT01253161/Prot_SAP_000.pdf